CLINICAL TRIAL: NCT05856305
Title: Phase II Randomized Study of Short Course Radiotherapy Based Total Neoadjuvant Therapy & Brachytherapy Boost With Or Without Chlorophyllin In Watch And Wait Suitable Locally Advanced Rectal Cancer (SCOTCH Study)
Brief Title: SCRT in TNT With or Without Chlorophyllin
Acronym: SCOTCH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 900959
Record Dates: First submitted 2023-04-10; First posted 2023-05-12 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-04

CONDITIONS: Rectal Neoplasms
Keywords: Locally Advanced rectal cancer; Sodium Copper Chlorophyllin
MeSH Terms: conditions — Rectal Neoplasms | interventions — chlorophyllin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorophyllin (Experimental): Drug name: Sodium Copper Chlorophyllin Dosage form: Tablet Dosage: 750 mg Route of administration: Oral Frequency: Once daily in the morning before food. Duration: From 10-14 days before radiotherapy up to 3 months after the last dose of cytotoxic therapy
  Interventions: Drug: Chlorophyllin, Sodium Copper Complex
- Placebo (Placebo Comparator): Drug Name: Placebo Dosage form: 1 Tablet Route of administration: Oral Frequency: Once daily in the morning before food. Duration: From 10-14 days before radiotherapy up to 3 months after the last dose of cytotoxic therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chlorophyllin, Sodium Copper Complex — Additional Chlorophyllin tablet with Short Course radiotherapy based total neoadjuvant treatment +/- brachytherapy boost dose
  Arms: Chlorophyllin
Drug: Placebo — Additional Placebo tablet with Short Course radiotherapy based total neoadjuvant treatment +/- brachytherapy boost dose
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to see, if addition of chlorophyllin to neoadjuvant Chemo-radiotherapy can reduce the gastro-intestinal/genitourinary/hematological toxicity rates and improve the quality of life in patient's diagnosed with locally advanced rectal cancer.

This is a randomized placebo control trial, wherein participants randomized to Chlorophyllin arm will receive the drug of interest along with the standard treatment. Participants randomized to other arm will receive placebo along with the standard treatment.

Researchers will compare the difference between the outcomes from both the arms and will also observe the non-operative management success rates.

DETAILED DESCRIPTION:
The current standard treatment for locally advanced rectal cancer includes neoadjuvant (treatment given before Surgery) radiotherapy & chemotherapy followed by surgery if needed or wait and watch in patients whom tumour has completely regressed. It has been observed that even after receiving this intensive treatment patients, almost 70% of patients develop acute toxicity (during or within 3 months) of grade 2 or higher (needing medication for toxicity). This affects their treatment tolerance, completion and quality of life.

In this study Researchers are going to see if addition of drug Chlorophyllin (derived from green plant leaves) along with standard treatment would help in reducing the acute toxicity. Chlorophyllin is present in all green leaves of plants giving them green color. The drug is derived from green plant leaves. As it is a plant-based product it is safe for humans and has no known side effects of its own. This is a randomized study which has two arms; Arm 1 is test arm where participants will receive drug of interest (Chlorophyllin) and in other arm participants will receive Placebo. Upon successful completion of study, outcomes from both the study arm will be compared and participants will be followed by standard protocol for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Histologically confirmed diagnosis of adenocarcinoma of the rectum.
* Clinical Stage II/III (T2-3, 4b: adherent to prostate, SV or post vagina but not grossly invading, N0-2) based on MRI.
* Non-circumferential tumours with craniocaudal length <7 cm
* The tumours of the lower rectum, or starting up to 7 cm from the anal verge.
* No evidence of distant metastases on CT Chest and Abdomen.
* No prior pelvic radiation therapy
* No prior chemotherapy or surgery for rectal cancer
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2
* Patients must read, agree to, and sign a statement of Informed Consent prior to participation in this study.
* Eligible to receive one of the options of standard neoadjuvant chemotherapy as determined by the medical oncologist team.

  * Absolute neutrophil count (ANC) > 1.5 cells/mm3, hemoglobin (HGB) > 8.0 gm/dl, platelet (PLT) > 150,000/mm3.
  * Total bilirubin ≤ 1.5 x ULN (except in patients with Gilbert's Syndrome who must have total bilirubin ≤ 3.0 x ULN), aspartate aminotransferase (AST) ≤ 3 x ULN, alanine transaminase (ALT) ≤ 3 x ULN.

Exclusion Criteria:

* Signet or mucinous histology cancer of rectum
* Recurrent rectal cancer or previous pelvic radiotherapy
* Primary unresectable rectal cancer.
* Creatinine level greater than 1.5 times the upper limit of normal.
* Patients who are unable to undergo an MRI.
* Patients with a history of any arterial thrombotic event within the past 6 months. This includes angina (stable or unstable), MI, TIA, or CVA.
* Ulcerative colitis or any other histologically confirmed inflammatory bowel disease.
* Patients with a history of venous thrombotic episodes such as deep venous thrombosis, and pulmonary embolism occurring more than 6 months prior to enrollment may be considered for protocol participation, provided they are on stable doses of anticoagulant therapy. Similarly, patients who are anticoagulated for a trial fibrillation or other conditions may participate, provided they are on stable doses of anticoagulant therapy.
* Patients with any other concurrent medical or psychiatric condition or disease which, in the investigator's judgment, would make them inappropriate candidates for entry into this study.
* Poor reliability for follow up.
* Ineligible as per eligibility criteria

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2027-09-09 (Estimated)

PRIMARY OUTCOMES:
Acute Toxicity | 3 months post-last cytotoxic therapy.
  Incidence of grade 2 or higher Common Terminology Criteria for Adverse Events (CTCAE) acute gastro-intestinal (GI)/genitourinary (GI)/haematological toxicity (HT) in advanced rectal cancer.
  Minimum value: Grade 1 Maximum value: Grade 5 Grade 1 late toxicity means a good outcome. Grade 2 or higher late toxicity means a worse outcome.

SECONDARY OUTCOMES:
Overall successful complete response rates | 3 years
  To estimate the 3-year overall complete response rates (clinical or pathological) and complete clinical response (cCR) at 24-36 weeks post TNT in whole cohort and if any difference between chlorophyllin and control arms.
Organ preservation rates | 3 years
  To estimate the 3-year organ preservation rates, TME free survival and if any difference between chlorophyllin & control arms.(by estimating patients who did not need surgery for rectal cancer (Total mesorectal excision; TME) at two years and if any difference between chlorophyllin and control arms.)
Disease free survival | 3 years
  To estimate the 3-year disease free survival, Distant metastasis free survival, loco-regional failure free survival, and overall survival rates in the whole cohort, and if any difference between two arms and between patients with successful non-operative management versus others.
Treatment related early and late toxicities | 2 years
  To compare treatment-related early and late toxicities (grade 2 Common Terminology Criteria for Adverse Events, version 5.0) for two years between the groups as (3).
  Minimum value: Grade 1 Maximum value: Grade 5 Grade 1 late toxicity means a good outcome. Grade 2 or higher late toxicity means a worse outcome.
Estimation of surgical complications | 30 days post surgery
  To estimate surgical complications based on Clavien-Dindo classification. Minimum value: Grade 1 Maximum value: Grade 5 Grade 1 surgical complications means a good outcome. Grade 2 or higher surgical complications means a worse outcome.
Health related quality of life | 2 years
  To estimate and compare Health Related Quality of Life (QOL) between various groups as (3). (using quality of life questionnaires (QLQ) of European Organization for Research and Treatment of Cancer (EORTC)) These questionnaires will be filled by patient at six month interval of follow up.
Cost benefit with reduction in toxicity | 2 years
  The direct cost of per patient for various supportive medications, hospital admissions will be estimated in both arms and compared to see if any financial benefit of reduction in toxicity.
  Record of medicines and details of hospitalization will be maintained.
Tumor Volume reduction kinetics | 2 years
  To study the correlation of tumour volume with used radiotherapy doses leading to a successful non-operative management versus not in the study group of patients.
To evaluate the timeline of Occurence | 3 years
  To evaluate the timeline of Occurence of grade 2/3 GI toxicities (namely rectal bleeding, rectal ulcer, rectal pain, tenesmus) during SCRT based TNT.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Rahul Krishnatry, M.D., Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No